CLINICAL TRIAL: NCT03981848
Title: Radiomics-based Non-invasive Classifier Research for HCC-related Liver Transplantation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zhejiang University (Other)
Collaborators: Fudan University (Other)
Responsible Party: Principal Investigator, Xiao Xu, professor, Zhejiang University
Other Study IDs: 2019ZJUXX-001
Record Dates: First submitted 2019-06-10; First posted 2019-06-11 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Hepatocellular Carcinoma; Liver Transplantation; Magnetic Resonance Imaging
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Relapse: Relapse of tumor within two years after liver transplantation
  Interventions: Other: Risk model of tumor relapse
- Non-relapse: Non-relapse of tumor within two years after liver transplantation
  Interventions: Other: Risk model of tumor relapse

INTERVENTIONS:
Other: Risk model of tumor relapse — High risk factor model of tumor relapse after liver transplantation
  Other Names: Risk model

SUMMARY:
The purpose of this study is to establish a non-invasive radiomics method to filter high recurrent-risk liver transplantation recipient population

DETAILED DESCRIPTION:
Hepatocellular carcinoma is one of the most common malignant tumors in the world with high incidence and mortality. Liver transplantation is the most effective treatment for HCC and is in high demand in China. However, recurrence of HCC among liver transplantation recipients is still a great challenge and threat to the survival of recipients. So it is of great significance to establish a non-invasive way to filter high liver transplantation recipient population before transplantation. Based on large scales of pre-treatment MR images, the investigator's study aims to establish a non-invasive radiomics method to filter high recurrent-risk liver transplantation recipient population. This study will contribute to the precise selection of HCC-related liver transplantation recipients.

ELIGIBILITY:
Inclusion Criteria:

* All patients had postoperative pathological diagnosis of HCC
* All patients had underwent contrast-enhanced MRI scan within 2 weeks before liver transplantation

Exclusion Criteria:

* patients whose pathological diagnosis is not HCC
* patients whose CT images were affected by strong imaging artifacts, i.e. artifacts obscuring more than 10% of whole volume of interest
* patients whose clinical data or CT images were missing

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospitalization patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
tumor recurrent status | two years